CLINICAL TRIAL: NCT07213960
Title: A Sequential Phase 2/3, Single-Arm, Open-Label Study in Adults Followed by a Randomized, Placebo-Controlled, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of APL2 in Adults and Adolescents With Focal Segmental Glomerulosclerosis
Brief Title: A Sequential Phase 2/3 Study of APL2 in Patients With Focal Segmental Glomerulosclerosis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APL2-FSG-319
Record Dates: First submitted 2025-09-15; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: FSGS
Keywords: Glomerulosclerosis; Focal Segmental; Child; Adult; Peptides; Cyclic; Complement Inactivator Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 2 - APL2 (Experimental): Sub-cutaneous infusions of APL2 (1080 mg / 20mL) twice weekly
  Interventions: Drug: APL2
- Phase 3 - APL2 (Experimental): Adults: Sub-cutaneous infusions of APL2 (1080 mg / 20mL) twice weekly
  Adolescents:
  ≥50 Kg: Sub-cutaneous infusions of APL2 (1080 mg / 20mL) twice weekly 35 to <50kg: First sub-cutaneous infusion of 648mg (12 mL) followed by 810mg (15 mL) every infusion thereafter (i.e. twice weekly) 30 to <35kg: First & Second sub-cutaneous infusion of 540mg (10mL) followed by 648mg (12 mL) every infusion thereafter (twice weekly)
  Interventions: Drug: APL2
- Phase 3 - Placebo (Placebo Comparator): Subcutaneous infusions of a sterile solution, twice-weekly, and equivalent in volume to the active arm based on participant's age and weight
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: APL2 — Complement (C3) Inhibitor
  Arms: Phase 2 - APL2; Phase 3 - APL2
Other: Placebo — Sterile solution of equal volume to active arm
  Arms: Phase 3 - Placebo

SUMMARY:
This is a sequential phase 2/3 study to evaluate the efficacy and safety of twice-weekly subcutaneous (SC) infusions of APL2 in patients diagnosed with FSGS. The initial phase 2 portion is a single-arm, open-label study in adults diagnosed with FSGS. Phase 2 will commence prior to randomizing for phase 3. The phase 3 portion of the study is a randomized, placebo-controlled, double-blinded, multicenter study in adults and adolescents diagnosed with FSGS.

ELIGIBILITY:
Inclusion Criteria:

* Age

  * Phase 2: adults aged ≥18 years
  * Phase 3: adults aged ≥18 years; if and where approved, adolescents (aged 12--17 years) at the time of signing the informed consent and assent form
* Weight ≥30 kg and ≤100 kg at screening
* FSGS diagnosis

  * Phase 2: primary, genetic, or undetermined FSGS diagnosed by kidney biopsy
  * Phase 3: primary, genetic, or undetermined FSGS diagnosed by kidney biopsy or by recognized podocyte genetic mutation
* At least 1.5 g/day of proteinuria on a screening 24-hour urine collection and a uPCR of at least 1.5 g/g in at least 2 FMU samples collected during screening
* Estimated glomerular filtration rate (eGFR) ≥25 mL/min/1.73 m2
* Stable regimen for FSGS treatment for at least 12 weeks prior to randomization, with no planned or anticipated adjustments or dose changes to the stable treatment regimen

Exclusion Criteria:

* Previous exposure to APL2
* Evidence of improving kidney disease in the 8 weeks prior to screening or during the screening period according to available data
* FSGS secondary to another condition (eg, infectious, diabetic, drug-induced, obesity, prematurity, sickle-cell, vesicoureteral reflux, congenital anomalies of the kidney, and urinary tract)
* Type 1 or uncontrolled (HbA1C ≥8%) type 2 diabetes mellitus
* History of kidney transplant
* Current or prior diagnosis of HIV, hepatitis B, or hepatitis C infection or positive serology or viral load during screening that is indicative of active infection with any of these viruses
* Hypersensitivity to APL2 or to any of the excipients
* Significant other kidney disease that would, in the opinion of the investigator, confound interpretation of study results
* Use of rituximab, belimumab, or any approved or investigational anticomplement therapy within 5 half-lives of that product prior to the screening period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Evaluate the efficacy of APL2 in terms of change from baseline in log-transformed urine protein to creatinine ratio (uPCR) | Baseline to Week 12
  Change from Baseline in Log-Transformed uPCR will be based on triplicate first morning urine (FMU)
Phase 3: Change from baseline in log-transformed urine protein to creatinine ratio (uPCR) | Baseline to Week 52
  Change from baseline in log-transformed uPCR will be based on triplicate first morning urine (FMU)

SECONDARY OUTCOMES:
Phase 2: Evaluate the efficacy of APL2 in terms of change from baseline in log-transformed urine albumin to creatinine ratio (uACR) | Baseline to Week 12
  Change From Baseline in Log-Transformed uACR will be based on first morning urine (FMU)
Phase 3: Change from Baseline in log-transformed urine protein to creatinine ratio (uPCR) | Baseline to Week 104
  Change from baseline in log-transformed uPCR will be based on triplicate first morning urine (FMU)
Phase 3: Proportion of participants achieving Complete Remission | Week 104
  Complete Remission is defined as participants who have achieved uPCR <0.3 g/g
Phase 3: Slope of estimated Glomerular Filtration Rate (eGFR) | Baseline to Week 104
  The annualized eGFR slope

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Investigator Site 1, Chicago, Illinois
  - Investigator Site 2, New York, New York